CLINICAL TRIAL: NCT03502967
Title: Imaging of Traumatic Brain Injury Metabolism Using Hyperpolarized Carbon-13 Pyruvate
Acronym: HPTBI
Status: Enrolling by invitation | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Jae Mo Park, Principal Investigator, University of Texas Southwestern Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: STU 072017-009
Record Dates: First submitted 2018-04-11; First posted 2018-04-19 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic Brain Injury; TBI
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Pyruvic Acid

STUDY DESIGN:
Intervention Model Description: TBI patients and healthy control subjects
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hyperpolarized [1-13C] Pyruvate (Experimental): Injection with hyperpolarized [1-13C] Pyruvate during MRI.
  Interventions: Drug: Hyperpolarized [1-13C] Pyruvate
- Hyperpolarized [2-13C] Pyruvate (Experimental): Injection with hyperpolarized [2-13C] Pyruvate during MRI.
  Interventions: Drug: Hyperpolarized [2-13C] Pyruvate

INTERVENTIONS:
Drug: Hyperpolarized [1-13C] Pyruvate — Bolus injection of study drug
  Other Names: HP Pyruvate Injection
  Arms: Hyperpolarized [1-13C] Pyruvate
Drug: Hyperpolarized [2-13C] Pyruvate — Bolus injection of study drug
  Other Names: HP Pyruvate Injection
  Arms: Hyperpolarized [2-13C] Pyruvate

SUMMARY:
This project is to evaluate sensitivity and specificity of hyperpolarized 13C-pyruvate as imaging agents of altered cerebral glycolysis and mitochondrial dysfunction and assess pyruvate utilization in mitochondria in Traumatic Brain Injury (TBI) patients.

DETAILED DESCRIPTION:
Aim 1:

Investigators will quantify changes in [1-13C]lactate and H13CO3- labeling following a bolus injection of hyperpolarized [1-13C]pyruvate during the time window of secondary injury to assess upregulated glycolysis. Due to heterogeneous presence and severity of damage by TBI, defining the injured brain region can be difficult. Therefore, the metabolite ratio maps ([product]/[pyruvate]) of TBI patients (n = 5) will be compared with those of healthy-controls (n = 3).

Hyperpolarized [2-13C]pyruvate will be examined in a separate group of TBI cohorts (n = 5) and healthy controls (n = 3), and [5-13C]glutamate, [1-13C]acetyl-carnitine, [1-13C]acetoacetate, and [1-13C]citrate from [2-13C]pyruvate will be quantified for assessing the altered mitochondrial metabolism. Imaging procedure with [2-13C]pyruvate is the same as the imaging with hyperpolarized [1-13C]pyruvate.

For both [1-13C]pyruvate and [2-13C]pyruvate studies, each subject will be imaged twice with a 45min interval for confirming the reproducibility of the methods and/or averaging to enhance the signal-to-noise ratios of 13C-metabolite maps.

Aim 2:

After the feasibility study (aim1) is completed, an intra-subject comparison study of [1-13C]pyruvate and [2-13C]pyruvate will be performed. Similar to the aim1, patients with post-TBI neurological disorders having normal or near-normal CT results (n = 6 patients) as well as normal brains of age/gender-matching healthy volunteers (n = 3) will be recruited. Each patient will be imaged twice (one with [1-13C]pyruvate and one with [2-13C]pyruvate with a 45min interval). PDH activity and the TCA cycling will be assessed from measured H13CO3- from hyperpolarized [1-13C]pyruvate and [5-13C]glutamate from [2-13C]pyruvate, respectively. The comparison of [1-13C]pyruvate and [2-13C]pyruvate will identify the detailed information of how pyruvate (and converted acetyl-CoA) is utilized in the mitochondria, and assess the utility and necessity of imaging hyperpolarized [2-13C]pyruvate in TBI, providing critical data for future grant applications and larger clinical trials.

ELIGIBILITY:
Inclusion Criteria:

TBI Patients

* Injury occurred within 30 days
* Documented and verified TBI by Glascow coma scal 10-15 and/or Loss of Consciousness >10 minutes.
* Head Computed Tomography at admission.

ALL Subjects:

* 18 through 60 years of age.
* Ability to understand the the willingness to sign a writteninformed consent.
* All races and ethnicities will be included; subjects must be able to read and speak either the English or Spanish language.

Exclusion Criteria:

* Non-traumatic structural brain abnormality identified on head CT.
* Metallic foreign bodies on the scalp or cranium which may interfere with MRI acquisitions.
* Penetrating TBI.
* Significant anatomic distortion of the brain identified on CT images, such as large hematomas, herniation, intraventricular hemorrhage, extensive subarachnoid hemorrhage, hydrocephalus.
* Significant polytrauma that would interfere with follow-up and outcome assessment.
* Patients on psychiatric hold.
* Major debilitating mental health disorders including, but not limited to schizophrenia and bipolar disorder that would limit compliance with study requirements.
* Major debilitating neurological disease including, but not limited to, stroke, CVA, dementia and tumor that would limit compliance with study requirements.
* Under influence of illicit drugs which are known to alter brain physiology/metabolism including, but not limited to cocaine, lysergic acid diethylamide (LSD), and marijuana at the time of MRI/MRSI scanning.
* Any contraindication per MRI Screening Form including
* Implants contraindicated at 3T, pacemakers
* Implantable Cardioverter Defibrillator (ICD)
* Claustrophobia
* Prisoners or patients in custody.
* Medically unstable including
* Heart failure
* Severe left ventricular outflow tract (LVOT) obstruction
* Unstable angina
* Pregnancy
* Lactating
* Subjects who are receiving any other investigational agents.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
[1-13C]lactate-to-H13CO3- ratio from [1-13C]pyruvate or [2-13C]lactate-to-[5-13C]glutamate ratio from [2-13C]pyruvate | One visit of three hours: 2 bolus injections during MRI with 45 minute rest period between the two
  Product ratio maps of lactate from pyruvate in the brain of TBI patients as compared to those of healthy controls.

CONTACTS AND LOCATIONS:
Locations (1):
- UT Southwestern - Advanced Imaging Research Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No